CLINICAL TRIAL: NCT00448123
Title: The Efficacy of Tamsulosin in the Treatment of Ureteral Stones in Emergency Department Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Swor (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Robert Swor, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-107
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Kidney Stones; Ureteral Stones
Keywords: Kidney Stones; Ureteral Stones; Flomax; Emergency Medicine; Urology
MeSH Terms: conditions — Kidney Calculi | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Tamsulosin (Active Comparator): Intervention - Tamsulosin
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin — Study Drug
  Other Names: Flomax
  Arms: Tamsulosin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To determine if emergency department patients with acute ureteral colic pain due to a ureteral stone who are treated with tamsulosin, versus placebo, will experience a shorter time to passage of their stone or resolution of their pain. A secondary study objective will be to determine if there is a relationship between response to tamsulosin and stone size or position in the ureter.

DETAILED DESCRIPTION:
This is a prospective randomized placebo controlled study of tamsulosin alone, vs placebo, to determine its effect on the rates of stone passage and resolution of pain in patients with acute renal colic pain that present to the emergency department. The study will be conducted in the Emergency Department (ED)and Emergency Department Observation Unit (EDOU) of William Beaumont Hospital, a high volume, university affiliated 952 bed suburban teaching hospital.

Patients will be given a seven-day supply of tamsulosin (0.4mg daily) or placebo. They will also be given a prescription for Vicodin (30 pills) and Ibuprofen (600mg, 30 pills). They will be called on days 1, 2, 3, 7, and 10 following the index visit regarding passage of stone or 48 hours without pain. Patients will be asked to call in if they pass their stone or are without pain for 48 hours. Related return visits to Royal Oak or Troy Beaumont within 30 days of their index visit will be followed by chart review.

The study will be limited to patients presenting to the emergency department with acutely symptomatic renal colic pain. Confirmation of a symptomatic stone will be made by imaging (helical CT scan or intravenous pyelogram).

Study exclusion criteria:

* Stone not documented on imaging
* Stones >10mm
* Pregnancy
* Age <18 years
* Evidence of infection with an obstructing stone
* Obstructing stone in a solitary kidney
* Currently taking tamsulosin, vardenafil, nifedipine, or steroids
* Contraindications or allergy to tamsulosin
* Ureteral surgery
* Patients that are unable to understand consent
* Patients that are unable to comply with follow-up

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department patients with acutely symptomatic renal colic pain
* Confirmation of a symptomatic stone will be made by imaging (helical CT scan or intravenous pyelogram).

Exclusion Criteria:

* Stones not documented on imaging
* Stones >10mm
* Pregnancy
* Age <18 years
* Evidence of infection with an obstructing stone
* Obstructing stone in a solitary kidney
* Currently taking tamsulosin, vardenafil, nifedipine, or steroids
* Contraindications or allergy to tamsulosin
* Ureteral surgery
* Patients that are unable to understand consent
* Patients that are unable to comply with follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2007-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Swor Robert, DO, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berger DA, Ross MA, Hollander JB, Ziadeh J, Chen C, Jackson RE, Swor RA. Tamsulosin does not increase 1-week passage rate of ureteral stones in ED patients. Am J Emerg Med. 2015 Dec;33(12):1721-4. doi: 10.1016/j.ajem.2015.08.006. Epub 2015 Aug 7. PMID 26429522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 127 subjects were enrolled in the study and 100 completed the study. Of the 27 that were excluded from analysis, 15 were excluded due to 'lost to follow-up', and another 12 had their stone removed surgically (physician decision) by the 7th day.
Groups:
- Placebo: None active placebo orally per day for up to 10 days.
- Tamsulosin: Tamsulosin orally 0.4 mg/daily for up to 10 days.
Period: Overall Study
Arm/Group | Placebo | Tamsulosin
Started | 62 | 65
Completed | 47 | 53
Not Completed | 15 | 12
Not completed — Lost to Follow-up | 9 | 6
Not completed — Physician Decision | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo Group
- Total: Total of all reporting groups
Arm/Group | Placebo | Tamsulosin | Total
Number analyzed (Participants) | 62 | 65 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 65 | 127
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 39 | 42 | 81
Region of Enrollment [Number; unit: participants]
  United States | 62 | 65 | 127

OUTCOME MEASURES:

1. Primary Outcome: Stone Passage
Description: Participants were asked during the follow-up phone call to indicate if their stone had passed within seven days. Phone calls were conducted at days 1, 2, 3, 7, 10 and 30 days after the emergency department discharge. Data is reported based on the information obtained up to the 7th day.
Time Frame: 1-7 days
Population: In the placebo group, of the 47 subjects 18 (46.2%) passed their stone by Day 7. In the Tamsulosin group, of the 53 subjects 21 (53.9%) passed their stone by Day 7.
Measure: Number; unit: participants
Arm/Group | Placebo | Tamsulosin
Number analyzed (Participants) | 47 | 53
participants | 18 | 21

2. Secondary Outcome: Amount (Mean Number of Tablets Taken) of Pain Medication Taken by Subjects up to Seven (7) Days Post Emergency Department Discharge
Time Frame: 1-7 days
Population: The data table is limited to the information collected at Day 7. Of the 53 subjects in the placebo group only 29 provided information regarding pain medication at the Day 7 interview. For the Tamsulosin group, only 15 out of 47 provided the pain medication information at the Day 7 interview. At Day 7 each group had only 3 non-zero responses.
Measure: Mean (Full Range); unit: Pain tablets
Groups:
- Placebo: Active placebo orally per day for up to 10 days.
Arm/Group | Placebo | Tamsulosin
Number analyzed (Participants) | 29 | 15
Pain tablets | 0.4 [0 to 4] | 0.6 [0 to 6]

3. Secondary Outcome: High Pain Score by Treatment Group
Description: Severity of Patient Pain at 7 days Post Emergency Department Visit. Patients were asked to describe their pain severity at each followup phone call, using a numerical scale, ranging from 0 (no pain) to 10 (worst possible pain). We report this measure at 7 days.
Time Frame: 7 Days
Population: The data table is limited to the information collected at Day 7. Of the 53 subjects in the placebo group only 29 provided information at the Day 7 interview. For the Tamsulosin group, only 15 out of 47 provided information at the Day 7 interview.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Placebo | Tamsulosin
Number analyzed (Participants) | 29 | 15
units on a scale | 1.69 [0 to 7] | 2.4 [0 to 8]

ADVERSE EVENTS:
Arm/Group | Placebo | Tamsulosin
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/53
Other Adverse Events (participants affected / at risk) | 5/47 | 4/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=47) | Tamsulosin (N=53)
Dizziness (Nervous system disorders) | 5 | 4

LIMITATIONS AND CAVEATS:
Limitations of this study include non-consecutive enrollment and small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes